CLINICAL TRIAL: NCT02402361
Title: Understanding Risk Factors and Determinants for Neuropathic Pain
Acronym: Neuropathic
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: Neuropathic Pain_DM_CTIL
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Diabetic Neuropathy
Keywords: Neuropathic pain; Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Understanding risk factors and determinants for neuropathic pain.

DETAILED DESCRIPTION:
Neuropathic pain (NP) is common (population prevalence of 7-8%) and will present a rising health burden in the future. NP arises as a consequence of a disease or lesion in the somatosensory nervous system. NP results in significant morbidity, reduces quality of life and has a major deleterious impact on health in aging. However, not everyone with such a lesion develops significant neuropathic pain, and those who do develop it include a wide range of severity, impact and outcomes, and an unpredictable response to evidence-based treatment. The reason why some subjects develop neuropathic pain and others do not following the same injury is not known. Genetic variants are increasingly recognized as being important in the development of neuropathic pain. There are a number of Mendelian primary neuropathic pain disorders which act as exemplars of high impact gene variants which have in a number of cases been shown to alter primary afferent excitability. In addition genetic factors are also likely to be important as risk factors in more common acquired (or secondary) neuropathic pain disorders. So, identifying these risk factors will have a significant impact on health both in identifying vulnerable patients and potential for developing new treatment modalities. The proposed study is a part of multicenter international project under Horizons 2020 program of the European Union. Our aim is to understand pain pathophysiology in terms of risk factors and protective mechanisms ranging from molecular pathways to societal impacts. The desired impact is to provide a firm platform to improve diagnosis and stratify patients according to risk profile, employ preventive strategies and ultimately develop novel therapeutics.

Specific objectives for the study at large will be to: 1) Identify the influence of demographic, environmental/societal and clinical factors on the risk of developing and maintenance of NP. 2) To apply modern genomics to validate (using a targeted approach) and find novel (using genome wide association) genetic risk factors for NP. 3) To determine if patient stratification using physiological (sensory profile, endogenous analgesic mechanisms and nerve excitability) and psychological factors can predict NP risk and progression. 4) Development of a risk model/algorithm for (severe) NP, combining measurable genetic and environmental factors. The desired impact is to provide a firm platform to improve diagnosis and stratify patients according to risk profile, employ preventive strategies and ultimately develop novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes who are ≥18 years of age who have a diagnosis of peripheral neuropathy based on a prior clinical assessment combined with supportive clinical investigations such as abnormal nerve conduction studies, reduced intraepidermal nerve or abnormal findings on quantitative sensory testing.
* If supportive clinical investigations (as described above) are not available at entry into the study, a neuropathy disability scale ≥3 will be required.
* Patients with symptoms highly suggestive of neuropathy that in the judgment of the clinical researcher are suitable for the study even if they do not fulfill other inclusion criteria.

Exclusion Criteria:

* Subjects who are pregnant.
* Subjects with insufficient command of Hebrew to obtain consent from or to complete the study questionnaires.
* Subjects with insufficient mental capacity to obtain consent from or complete study questionnaires.
* Subjects with concurrent severe psychological or psychiatric disorders.
* Patients with moderate to severe pain form other causes that may confound assessment or reporting of pain.
* Patients with central nervous lesions, which may complicate somatosensory testing.
* Who is in the opinion of the investigator unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients with painful and non-painful diabetic neuropathy (males and females, ages ≥18) will be tested in the study performed in the Rambam Medical Center. The patients will be recruited from the neurology/diabetes clinics and by advertisement in local newspapers.
  No patients will be requested to withdraw from any of their medication, or to change the treatment regimen due to participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Risk factors and determinants for neuropathic pain | 4 years
  Identify the influence of demographic, environmental/societal and clinical factors on the risk of developing and maintenance of NP

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Topaz LS, Frid A, Granovsky Y, Zubidat R, Crystal S, Buxbaum C, Bosak N, Hadad R, Domany E, Alon T, Meir Yalon L, Shor M, Khamaisi M, Hochberg I, Yarovinsky N, Volkovich Z, Bennett DL, Yarnitsky D. Electroencephalography functional connectivity-A biomarker for painful polyneuropathy. Eur J Neurol. 2023 Jan;30(1):204-214. doi: 10.1111/ene.15575. Epub 2022 Oct 26. PMID 36148823